CLINICAL TRIAL: NCT00578617
Title: Catheter Ablation Versus Antiarrhythmic Drug Therapy for Atrial Fibrillation - Pilot Trial
Brief Title: Ablation vs Drug Therapy for Atrial Fibrillation - Pilot Trial
Acronym: CABANA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Duke Clinical Research Institute (Other); Abbott Medical Devices (Industry)
Responsible Party: Douglas L. Packer, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-003867
Record Dates: First submitted 2007-12-14; First posted 2007-12-21 (Estimated); Results first posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2012-12

CONDITIONS: Atrial Fibrillation; Arrhythmia
Keywords: Atrial fibrillation; Left Atrial Ablation; Pulmonary Vein Isolation; Catheter Ablation; Antiarrhythmic Drug Therapy
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Heart Rate; Metoprolol; Atenolol; Propranolol; Acebutolol; Carvedilol; Diltiazem; Verapamil; Digoxin; Sotalol; Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pharmacologic Therapy (Active Comparator): Pharmacologic Therapy Rate and/or Sinus Rhythm Control: Patients without other heart disease will receive beta or calcium channel blockers as first line rate control therapy. Patients with underlying coronary artery disease will receive beta-blockers, patients with limited ventricular hypertrophy not warranting exclusion would receive either beta- or calcium channel blockers, while patients with heart failure would be expected to receive carvedilol or metoprolol. Patients randomized to drug therapy may be started on a membrane active drug, in an approach consistent with the recommended Guidelines for Management of Subjects with AF. Each patient will be placed on an anti-arrhythmic drug for an appropriate period and the patient cardioverted to sinus rhythm if necessary. Patients will then be followed for a period of up to 3 months, during which dosage adjustment can be made or the drug replaced with a different anti-arrhythmic drug.
  Interventions: Drug: Rate Control; Drug: Rhythm Control
- Ablation Therapy (Active Comparator): Left Atrial Catheter Ablation: The specific choice of ablation catheters will be left to the investigator from the following list: Lifewire TC XLS, Therapy Dual/Thermocouple, NAVI-STAR/NAVI-STAR DS, Celsius Braided Tip, NAVI-STAR Thermo-Cool, Freezor/FreezorMax, Stinger, Blazer II RF/RPM/SteeroCath /XP, Chilli Cooled.
  Interventions: Device: Ablation Therapy

INTERVENTIONS:
Drug: Rate Control — Metoprolol 50-100mg
  Other Names: Toprol
  Arms: Pharmacologic Therapy
Device: Ablation Therapy
  Other Names: St. Jude: Livewire
  Arms: Ablation Therapy
Drug: Rate Control — Atenolol 50-100mg,
  Other Names: Tenormin
  Arms: Pharmacologic Therapy
Drug: Rate control — Propranolol 40-80mg
  Other Names: Inderal
  Arms: Pharmacologic Therapy
Drug: Rate control — Acebutolol 200mg
  Other Names: Sectral
  Arms: Pharmacologic Therapy
Drug: Rate control — Carvedilol 6.25mg
  Other Names: Coreg
  Arms: Pharmacologic Therapy
Drug: Rate Control — Diltiazem 180-240mg
  Other Names: Cardizem
  Arms: Pharmacologic Therapy
Drug: Rate Control — Verapamil 180-240mg
  Other Names: Calan
  Arms: Pharmacologic Therapy
Drug: Rate Control — Digoxin 0.125mg
  Other Names: Lanoxin
  Arms: Pharmacologic Therapy
Drug: Rhythm Control — Propafenone 450mg
  Other Names: Rhythmol
  Arms: Pharmacologic Therapy
Drug: Rhythm control — Flecainide 200mg
  Other Names: Tambacor
  Arms: Pharmacologic Therapy
Drug: Rhythm control — Sotalol 240mg
  Other Names: Betapace
  Arms: Pharmacologic Therapy
Drug: Rhythm control — Dofetilide 500mcg
  Other Names: Tykosin
  Arms: Pharmacologic Therapy
Drug: Rhythm control — Amiodarone 200mg
  Other Names: Cordarone
  Arms: Pharmacologic Therapy
Drug: Rhythm control — Quinidine 600-900mg
  Other Names: Quini-glute/dex
  Arms: Pharmacologic Therapy

SUMMARY:
The CABANA pilot study is designed to test the hypothesis that the treatment strategy of percutaneous left atrial catheter ablation for the purpose of the elimination of atrial fibrillation (AF) is superior to current state-of-the-art therapy with either rate control or anti-arrhythmic drugs for reducing AF recurrences at 1 year follow-up.

DETAILED DESCRIPTION:
The need for this trial arises out of 1) the rapidly increasing number of pts > 60 years of age with AF accompanied by symptoms and morbidity, 2) the failure of anti-arrhythmic drug therapy to maintain sinus rhythm and reduce mortality, 3) the rapidly increasing application of radio-frequency catheter ablation without appropriate evidence-based validation, and 4) the expanding impact of AF on health care costs.

ELIGIBILITY:
Inclusion Criteria:

* Have documented AF, which warrants active drug or ablative treatment
* Be eligible for both catheter ablation and at least 2 sequential anti-arrhythmic drugs and/or 3 sequential rate control drugs
* Be >65 yrs of age, or <65 yrs with one or more of the following risk factors for stroke: Hypertension, Diabetes, Congestive heart failure (including systolic or diastolic heart failure), Prior stroke or transient ischemic attack, Left atrium >4.5 cm, ejection fraction <35% by echocardiogram, radionuclide evaluation or contrast ventriculography

Exclusion Criteria:

* Previously failed 2 or more membrane active anti-arrhythmic drugs
* Efficacy failure of a full dose Amiodarone trial of >12 weeks duration
* Any amiodarone therapy in the past three months
* Reversible causes of AF including thyroid disorders, acute alcohol intoxication, recent major surgical procedures, or trauma
* Lone atrial fibrillation in the absence of risk factors for stroke in patients <65 years of age
* Recent cardiac events including myocardial infarction, percutaneous intervention, or valve or coronary bypass surgery in the preceding 3 months
* Hypertrophic obstructive cardiomyopathy
* Class IV angina or congestive heart failure
* Planned heart transplantation
* Other mandated anti-arrhythmic drug therapy
* Heritable arrhythmias or increased risk for "torsade de pointes" (a specific, rare variety of ventricular tachycardia) with class I or III drugs
* Prior left atrial catheter ablation with the intention to treat AF
* Patients with other arrhythmias requiring ablative therapy
* Prior surgical interventions for AF such as the MAZE procedure
* Prior atrioventricular nodal ablation
* Medical conditions limiting expected survival to <1 year
* Contraindication to warfarin anti-coagulation
* Women of childbearing potential
* Participation in any other clinical mortality trial
* Unable to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-09; Primary Completion 2009-02 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas L. Packer, M.D., Principal Investigator — Mayo Clinic
Locations (10):
- United States (10):
  - Universtity of Alabama Hospital, Birminham, Alabama
  - Good Samaritan Hospital, Los Angeles, California
  - Loyola University, Maywood, Illinois
  - Mercy Medical Center, Des Moines, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Pennsylvania Health, Philadelphia, Pennsylvania
  - Intermountain Medical Center, Murray, Utah

REFERENCES:
- [Background] Cleland JG, Coletta AP, Buga L, Ahmed D, Clark AL. Clinical trials update from the American College of Cardiology meeting 2010: DOSE, ASPIRE, CONNECT, STICH, STOP-AF, CABANA, RACE II, EVEREST II, ACCORD, and NAVIGATOR. Eur J Heart Fail. 2010 Jun;12(6):623-9. doi: 10.1093/eurjhf/hfq083. PMID 20498271

RESULTS

PARTICIPANT FLOW:
Groups:
- Drug Therapy: Pharmacologic Therapy Rate and/or Rhythm Control: MD to choose from this list as medically indicated, doses are min recommended daily dose: metoprolol 50-100 mg, atenolol 50-100 mg, propanolol 40-80 mg, acebutolol 200 mg, carvedilol 6.25 mg, diltiazem 180-240 mg, verapamil 180-240 mg, digoxin 0.125 mg, propafenone 450 mg, flecainide 200 mg, sotalol 240 mg, dofetilide 500 mcg, amiodarone 200 mg, quinidine 600-900 mcg.
Period: Overall Study
Arm/Group | Drug Therapy | Ablation Therapy
Started | 31 | 29
Completed | 31 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug Therapy | Ablation Therapy | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 18 | 38
  >=65 years | 11 | 11 | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 62.1 (9.57) | 60.3 (11.46) | 61.2 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 26 | 20 | 46
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Recurrence of Atrial Fibrillation by One Year Follow-up
Description: Documentation of atrial fibrillation using a cardiac event recorder
Time Frame: 12 months after intervention
Measure: Number; unit: participants
Arm/Group | Drug Therapy | Ablation Therapy
Number analyzed (Participants) | 31 | 29
participants | 20 | 14

ADVERSE EVENTS:
Time Frame: Subjects were followed for adverse events for the 1 year they were on this trial.
Arm/Group | Drug Therapy | Ablation Therapy
Serious Adverse Events (participants affected / at risk) | 4/31 | 12/29
Other Adverse Events (participants affected / at risk) | 8/31 | 10/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Therapy (N=31) | Ablation Therapy (N=29)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (2) | 1 (2)
Adverse (General disorders) | 1 (1) | 0 (0)
Cardiac Tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Vascular Pseudoaneurysm (Vascular disorders) | 0 (0) | 1 (1)
Device Related Infection (Infections and infestations) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Coronary Artery Occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1)
Arteriovenous Fistula (Vascular disorders) | 0 (0) | 1 (1)
Ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Therapy (N=31) | Ablation Therapy (N=29)
Vascular Injury (Vascular disorders) | 1 (1) | 2 (2)
Haematoma (Vascular disorders) | 1 (1) | 2 (2)
Rash (General disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Transient Ischaemic Attack (Vascular disorders) | 0 (0) | 1 (1)
Fluid Overload (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Cardiac Failure (Cardiac disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
Limited number enrolled. Study was designed to demonstrate feasibility for a pivotal trial, but small enrollment limits the final conclusions that can be drawn from a simple 'time to first atrial fibrillation recurrence.'

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No